CLINICAL TRIAL: NCT00697307
Title: A Bioequivalence Study Of A Low Cumulative Release Lot Of Norelgestromin (NGMN)/Ethinyl Estradiol (EE) Transdermal Contraceptive Systems Compared With Currently Marketed Ortho-Evra In Healthy Female Volunteers
Brief Title: Bioequivalence Study of Patches With Different Release Profiles
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Other Study IDs: CR002626
Record Dates: First submitted 2008-06-05; First posted 2008-06-13 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Female Contraception
Keywords: bioequivalence; contraception; contraceptive patch; ORTHO EVRA; norelgestromin; NGMN; ethinyl estradiol; EE

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study was to determine the bioequivalence of a norelgestromin/ethinyl estradiol (NGMN/EE) transdermal contraceptive system.

DETAILED DESCRIPTION:
The primary objective was to determine the bioequivalence of a norelgestromin/ethinyl estradiol (NGMN/EE) transdermal contraceptive system lot with a cumulative release profile below the lower limit of the specifications (low spec lot) compared with a currently marketed lot of EVRANORELGESTROMIN/ETHINYL ESTRADIOL with a cumulative release profile well within the specifications limits (reference lot), after application to the buttock. This was a single center, randomized, double-blind, 2 way crossover study. The double-blind treatment phase included two 7-day treatment periods separated by a 28 day washout period. Safety was assessed throughout the study. The study population was comprised of healthy women aged 18 to 45 years, inclusive, who weighed at least 110 pounds with a body mass index (BMI) between 16 and 29.9 kg/m2, and a hematocrit of at least 36%. Eligible patient were randomly assigned to 1 of 2 treatment sequence groups. A 20 cm2 NGMN/EE transdermal contraceptive patch (low spec lot [test] or EVRANORELGESTROMIN/ETHINYL ESTRADIOL [reference]) was applied to each patient on the buttock and worn for 7 days. Twenty-eight days after removal of the first patch (Day 36 of Period 2), the patient crossed over to the other treatment. After each patch was removed, the skin was checked for redness and swelling. Blood samples were collected for measurement of drug concentrations during the 7-day wear periods and for 3 days after each patch was removed. Patients were telephoned weekly during the washout period to remind them to use back-up contraception. After the last blood sample collection on Day 46, or in instances where the patient withdrew early from the study, post treatment procedures including physical and gynecologic examinations, vital signs, laboratory evaluations, and a serum pregnancy test were performed. The following pharmacokinetic parameters were to be estimated for NGMN, NG, and EE after low spec lot and EVRANORELGESTROMIN/ETHINYL ESTRADIOL patch application: Cmax - maximum observed serum concentration after patch application; tmax - time of maximum serum concentration after patch application; Css - mean steady-state concentration for NGMN and EE after patch application calculated as the mean concentration between 48 and 168 hours; Cavg - average concentration for NG calculated as AUC168/168; AUC - the area under the serum concentration-time curve for NGMN, NG, and EE using linear trapezoidal summation from the data obtained after patch application from time 0 (dosing) to 168 hours post dose (AUC168), from time 0 to 240 hours postdose (AUC240), from time 0 to infinity (AUCinf), and from time 0 to the last measurable concentration for EE (AUClast); and t½ - apparent terminal half-life, computed as (ln2/ke) where ke is the slope of the terminal log-linear phase of the serum concentration-time curve. Patch adhesion was assessed and scores summarized. Assessment of bioequivalence will be based on the use of 90% confidence intervals (for 2 one-sided test procedures) for the ratios of mean (low spec lot to EVRANORELGESTROMIN/ETHINYL ESTRADIOL ) pharmacokinetic parameters, AUC240 and Css for NGMN and EE. The 2 formulations will be considered bioequivalent if the 90% confidence intervals fall within 80% to 125% limits for both AUC240 and Css for NGMN and EE. Safety evaluations were based on adverse events, including erythema and application site reaction and changes in physical and gynecologic examinations (including breast exams), vital signs, 12-lead ECGs, and clinical laboratory test results from pre- to poststudy. Serum pregnancy testing and urine drug screening was performed. Changes from screening were summarized using descriptive statistics. A single low spec lot or EVRANORELGESTROMIN/ETHINYL ESTRADIOL patch (20 cm2 transdermal contraceptive system) contains NGMN 6.0 mg and EE 0.75 mg. Each subject wore a patch (low spec lot or EVRANORELGESTROMIN/ETHINYL ESTRADIOL ) on the buttock for 7 days, according to a computer-generated randomization schedule. There was a 28-day washout period. Patients then crossed over to the other treatment for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by physical and gynecologic examinations, clinical laboratory assessments, vital sign measurements, and a 12-lead electrocardiogram (ECG)

Exclusion Criteria:

* Pregnant
* Lactating
* Currently using hormonal contraceptive

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2003-03; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Bioequivalence study of patches with different release profiles — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=482&filename=CR002626_CSR.pdf